CLINICAL TRIAL: NCT04450160
Title: A Phase 2, Randomized, Open-Label Study of Anhydrous Enol-Oxaloacetate in Subjects With Newly Diagnosed Glioblastoma Multiforme
Brief Title: Trial of AEO in New Glioblastoma (GBM)
Acronym: AEO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: MetVital, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Terra-001-201
Record Dates: First submitted 2020-06-23; First posted 2020-06-29 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Glioblastoma Multiforme
Keywords: Glioblastoma; Oxaloacetate; Seizures; Warburg
MeSH Terms: conditions — Glioblastoma; Seizures | interventions — Standard of Care; Drug Therapy; Temozolomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Placebo Comparator): Current GBM Treatment of surgery, radiation and chemotherapy with temozolomide.
  Interventions: Other: Standard of Care
- AEO with Standard of Care (Experimental): Anhydrous Enol-Oxaloacetate added to the Standard of Care (surgery, radiation and chemotherapy with temozolomide).
  Interventions: Drug: Anhydrous Enol-Oxaloacetate (AEO); Other: Standard of Care

INTERVENTIONS:
Drug: Anhydrous Enol-Oxaloacetate (AEO) — Oral supplementation with AEO along with the Standard of Care (Temozolomide)
  Arms: AEO with Standard of Care
Other: Standard of Care — Standard of Care Temozolomide
  Other Names: Chemotherapy with Temozolomide

SUMMARY:
This is a multicenter, Phase 2, Proof-of-concept study in subjects with newly diagnosed glioblastoma multiforme (GBM).

All subjects will receive standard of care therapy for the treatment of their GBM and any Anti-Epileptic Drug (AED) deemed necessary for their surgical resection of the GBM. Patients who are taking concomitant AEDs will be eligible for the study. Treatment with Anhydrous Enol-Oxaloacetate will be added to the Standard of Care.

This study is testing adjuvant Anhydrous Enol-Oxaloacetate (AEO) in GBM, an orally active drug candidate which in animal studies has demonstrated decreased tumor growth rate and increased survival.

DETAILED DESCRIPTION:
Currently, the multidisciplinary Standard of Care treatment for Glioblastoma multiforme includes maximal surgical resection of the tumor followed by radiotherapy plus concomitant and maintenance temozolomide chemotherapy.This study will treat newly diagnosed GBM patients by adding Anhydrous Enol-Oxaloacetate treatment to their current Standard of Care.

In the body, Anhydrous Enol-Oxaloacetate (AEO) converts into "Oxaloacetate", a metabolite important for many biochemical reactions in the body. On a cellular level, oxaloacetate treatment has been found to modify cancer metabolism in GBM cells, reversing the "Warburg Effect", reducing glycolysis and reducing lactate production. In animals, oxaloacetate treatment has increased survival and reduced tumor growth of implanted GBM tumors.

In other animal studies, oxaloacetate has also shown to have neuo-protective effects including positive effects on seizure development.

.

ELIGIBILITY:
Inclusion Criteria:

* • Histopathologic diagnosis of glioblastoma multiforme

  * Standard of care maximal feasible surgical resection of the glioma
  * Post-operative pre-enrollment MRI-Note: measurable disease is not required
  * Concomitant anti-epileptic drugs
  * Hemoglobin >9 g/dL
  * Platelets >100,000/microliter (mcL)
  * <3.0 Upper Limit of Normal Range (ULN) for Alanine aminotransferase (ALT), Aspartate aminotransferase (AST) and/or Alkaline Phosphatase
  * <2.0 Upper Limit of Normal Range (ULN) for serum creatinine
  * Karnofsky performance status >70
  * Mentally competent to follow study procedures
  * Male and female patients of childbearing potential must agree to use a dual method of contraception (a highly effective method of contraception in conjunction with barrier contraception) consistently and correctly from the first dose of study drug until 90 days after the last dose of study drug
  * Able to answer questions on the Patient-Reported Outcomes Measurement Information System (PROMIS) questionnaire
  * Subject is willing and able to give informed consent and to follow instructions as per the protocol

Exclusion Criteria:

* • Concomitant treatment with carmustine wafers or tumor-treating electric fields (TTFields)

  * QT Interval corrected with the fridericia formula (QTcF) >480ms
  * Significant concurrent illness / disease
  * Predicted life expectancy < 6 months from date of randomization
  * Pregnancy
  * Enrollment in another clinical trial during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 6 months
  Measurement of Overall Survival
Progression Free Survival-6 | 6 months
  Survival at 6 months

SECONDARY OUTCOMES:
Seizures | 6 months
  Time from randomization to first seizure
Chalfont-National Hospital Seizure Severity | 6 months
  Measure of Seizure Severity Ranging from a minimum of 1 to a maximum of 27 with higher score indicating worse outcome
PROMIS-Cancer - Fatigue | 6 months
  Measure of Fatigue Ranging from a minimum of 0 to a maximum of 95 with the higher score indicating worse outcome.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Augur ZM, Doyle CM, Li M, Mukherjee P, Seyfried TN. Nontoxic Targeting of Energy Metabolism in Preclinical VM-M3 Experimental Glioblastoma. Front Nutr. 2018 Oct 5;5:91. doi: 10.3389/fnut.2018.00091. eCollection 2018. PMID 30349820
- [Background] Ruban A, Berkutzki T, Cooper I, Mohar B, Teichberg VI. Blood glutamate scavengers prolong the survival of rats and mice with brain-implanted gliomas. Invest New Drugs. 2012 Dec;30(6):2226-35. doi: 10.1007/s10637-012-9799-5. PMID 22392507
- [Background] Yamamoto HA, Mohanan PV. Effect of alpha-ketoglutarate and oxaloacetate on brain mitochondrial DNA damage and seizures induced by kainic acid in mice. Toxicol Lett. 2003 Jul 20;143(2):115-22. doi: 10.1016/s0378-4274(03)00114-0. PMID 12749815